CLINICAL TRIAL: NCT04819685
Title: Application of KANG FU PEN (Protective Irrigation Solution Against Rays) in Radical Concurrent Radiotherapy and Chemotherapy for Cervical Cancer to Prevent and Treat Radiation-induced Rectal Injury：a Multicenter, Prospective, Randomized Trail
Brief Title: Application of KANG FU PEN in Radical Concurrent Radiotherapy and Chemotherapy for Cervical Cancer to Prevent and Treat Radiation-induced Rectal Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Chinese PLA General Hospital (Other); Peking University Third Hospital (Other); Peking University Cancer Hospital & Institute (Other); Jiangsu Cancer Institute & Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Sun Yat-sen University (Other); Jilin Provincial Tumor Hospital (Other); Fudan University (Other); Shandong Cancer Hospital and Institute (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Guizhou Cancer Hospital (The Affiliated Cancer Hospital of Guizhou Medical University) (Unknown); Zhejiang Cancer Hospital (Other); Xiangya Hospital of Central South University (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFP for RTI rectal injury
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer; Radiotherapy Side Effect; Radiotherapy; Complications
MeSH Terms: conditions — Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Intervention:Anti-radiation spray (liquid dressing)
  Interventions: Drug: KANG FU PEN
- control group (No Intervention)

INTERVENTIONS:
Drug: KANG FU PEN — FU PEN: anti-radiation spray (liquid dressing) treatment which is a protective irrigation solution against rays
  Arms: test group

SUMMARY:
A total of 520 cases will be randomly divided into Kang Fu Pen (liquid dressing) enema intervention group (experimental group) and non-enema intervention group (control group), according to the ratio of 1:1.

DETAILED DESCRIPTION:
All patients are planned to receive radical concurrent chemoradiotherapy. Intensity modulated radiotherapy (IMRT) will be used for external irradiation, with a dose of 45-50.4Gy /25-28 fractions. Combined three-dimensional intracavitary/interstitial (IC/IS) brachytherapy was applied. The preferred dose fraction plan is 6Gy*5 fractions, or 7Gy*4 fractions. Whether to adopt supplement radiotherapy can be decided by the tumor regression. Cisplatin 40 mg/m2 is recommended as the first choice for concurrent chemotherapy, and TP or TC can also be considered. Single-drug weekly therapy should be completed for at least 3 cycles, and combined 3-week regimen should be completed for at least 1 cycle.

Experimental group: from three days before radiotherapy to one week after radiotherapy, Kang Fu Pen (recombinant human superoxide dismutase) retention enema, 50ml/ time, once every other day. When rectal mucosa II degree reactions (NCI-CTCAE 5.0) occur, it is changed to 1 day/time until 1 week after mucosal remission.

Control group: 3 days before radiotherapy to the end of radiotherapy, no drug retention enema was used.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is completely voluntary and has the ability to sign the research informed consent form within 30 days before enrollment;
2. Age ≥18 years old and ≤65 years old;
3. Pathologically confirmed cervical cancer;
4. Those with IB3, IIA2, IIB, IIIA, IIIB, and those with cervical tumor ≥ 4cm or involved parametrial in IIIC1 and IIIC2 (FIGO 2018 staging);
5. ECOG score 0-2 points;
6. The complete blood count and basal metabolic indexes in the 14 days before enrollment must meet the following requirements: NEUT≥1.5*10^9/L, HGB≥80g/L, PLT≥100*10^9/L, blood creatinine < 1.5mg/dl (133umol/L), AST and ALT are within 2 times of the upper limit of normal;
7. Those who have had regular bowel movements and had a negative stool routine test + occult blood before enrollment.

Exclusion Criteria:

1. Those who have a history of allergy to superoxide dismutase use;
2. Patients with skin and mucous membrane infections, patients with obvious empyema or pelvic inflammatory disease;
3. Those who have had chronic colitis, ulcerative colitis, and non-specific proctitis in the past;
4. Those who have received cervical cancer surgery (including pelvic or retroperitoneal lymphadenectomy, excluding tumor biopsy), radiotherapy or chemotherapy;
5. Those who are expected to be unable to receive brachytherapy, or brachytherapy needs to use tumor elimination, uterine tube inserted alone in one fraction, or template plan;
6. Those who need to use fluorouracil or capecitabine or tigio in the concurrent chemotherapy regimen;
7. History of other malignant tumors;
8. Pregnant or lactating women;
9. Accompanied by active infection and fever;
10. Other serious diseases that may significantly affect the compliance of clinical trials, such as unstable heart disease, kidney disease, chronic hepatitis, poorly controlled diabetes, and mental illness that require treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Degree of rectal mucosal injury caused by acute radiation | Within 1 week after radiotherapy
  the incidence of Vienna rectoscopy score ≥2 within 1 week after radiotherapy. Vienna rectoscopy score was used.

SECONDARY OUTCOMES:
Degree of rectal injury caused by chronic radiation | 3 to 24 months after radiotherapy
  incidence of RTOG score ≥2 at 3 to 24 months after radiotherapy. If the RTOG score ≥2 at 3 to 24 months after radiotherapy, rectoscopy will be used to evaluate the degree. If the RTOG score is 0 or 1, clinical classification is enough.
Quality of life score | 3 to 24 months after radiotherapy
  EORTC QLQ-C30 (V3.0) was used to score quality of life before, during, and after radiotherapy.
overall survival (OS) | 3 years after radiotherapy
  Overall survival (OS) is defined as the time interval from randomization to death from any cause or, if no death, to the last follow-up.
disease-progression-free survival (PFS) | 3 years after radiotherapy
  Progression-free survival (PFS) is defined as the time between randomization and the occurrence of local or regional recurrence, or distant metastasis, or death from any cause, based on the time of the first event and, if none of these events occurred, to the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No